CLINICAL TRIAL: NCT06167382
Title: Acute Effect of Arm Ergometer Exercise Intensity on Dexterity and Hand Reaction Time
Brief Title: The Effect of Arm Ergometer Exercise on Dexterity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ArmErgometer
Record Dates: First submitted 2023-08-12; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-09

CONDITIONS: Healthy Adults; Upper Extremity; Dexterity
Keywords: Acute effect; Arm ergometer; Dexterity; Reaction time

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Female and Male Adults (Experimental): Demographic Survey Form,the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+),Digital Dynamometer Measurement,ROM Measurements, Muscle Strength Tests, Grip Strength Measurement, Hand Skill and Function Tests, Arm Ergometer,Modified Borg Scale, Pulseoximeter will be applied to the participants.
  Interventions: Other: Questionnare; Other: Device: Arm Ergometer

INTERVENTIONS:
Other: Questionnare — Demographic Survey Form,the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+),Goniometric Measurements, Digital Dynamometer Measurements, Hand Grip Measurements, Hand Reaction Measurements, Dexterity and Function Measurements, Jamar Handheld Dynomometer Measurement, Pinchmeter Measurement, Purdue Pegbord Test, Minnesota Manuel Skill Test, Nelson Hand Reaction Test, Modified Borg Scale
Other: Device: Arm Ergometer — Participants will sign a consent form approved by the ethics comittee. Before data collection height, weight, daily computer usage time, dominant hand, body mass index, heart rate, blood pressure and saturation values be recored. Before arm ergometer exercise, the muscle strength, hand grip strength, joint range of motion, dexterity and reaction speed will be evaluated. The dexterity and reaction speed will be done with Minnesota Manuel Skill Test, Purdue Pegbord Test and Nelson Hand Reaction Test.Participants will be training at least 24 hours apart at 60%, 70%, and 80% of exercise intensity maximum heart rate on arm ergometer. The tests will repeat at the same time with a maximum deviation of 1 hour on 3 different days. At the end of arm ergometer exercise, the necessary evaluations will be made again and the participants will be rest for 15 minutes. 15 minutes after the participants rested, the necessary evaluations will be made again.

SUMMARY:
The goal of this single group assessment study is to investigate acute effect of arm ergometer exercise intensity on dexterity and hand reaction time in healthy male or female participants aged 18-35.

* Knowing the acute effect and change of hand dexterity and reaction times of individuals with arm ergometer intensities applied at different intensities provides us with data that can be processed and used in neurological, orthopedic patient groups and geriatric cases during the rehabilitation process.
* The positive gains enable us to obtain effective and observable results in the rehabilitation progression of individuals and in parameters such as muscle strength and endurance, quality of life, depression, chronic pain.

Participants who accepted the voluntary basis will be taken and the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) will be filled. After all evaluations were made to the participants, 3 different exercise intensities; maximum heart rates; 60%, 70%, 80% will do arm ergometer exercises.

* ROM measurements
* Muscle strength tests
* Grip strength measurement (Jamar hand dynamometer)
* Dexterity and Function tests (Nelson Hand Reaction Test
* Purdue Pegboard Test
* Minnesota Manual Dexterity Test) evaluation parameters will be applied before, immediately after and 15 minutes after each exercise intervention.

DETAILED DESCRIPTION:
In this study on the acute effect of arm ergometer exercise intensity on dexterity and hand reaction time; Knowing the acute effect and change of hand dexterity and reaction times of individuals with arm ergometer intensities applied at different intensities provides us with data that can be processed and used in neurological, orthopedic patient groups and geriatric cases during the rehabilitation process. The positive gains enable us to obtain effective and observable results in the rehabilitation progression of individuals and in parameters such as muscle strength and endurance, quality of life, depression, chronic pain.

Arm ergometer exercise is an upper extremity aerobic exercise. Aerobic exercises are exercises that increase the capacity and efficiency of this system by using the cardiorespiratory system. In the literature; In addition to the small number of studies examining the acute effects of arm ergometer exercises, it is noteworthy that there is no consensus on the effect on dexterity and hand reaction time. In the literature review, no study was found that examined the effect of arm ergometer exercise at different intensities on dexterity and hand-eye coordination.

The aim of this study; To determine the effect of arm ergometer exercise intensity levels on dexterity and hand reaction time. On the basis of this study, demographic data of 23 healthy male or female participants aged 18-35, who accepted the voluntary basis, will be taken and the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) will be filled. After all evaluations were made to the participants, 3 different exercise intensities; maximum heart rates; 60%, 70%, 80% will do arm ergometer exercises. ROM measurements, Muscle strength tests, Grip strength measurement (Jamar hand dynamometer), Dexterity and Function tests (Nelson Hand Reaction Test, Purdue Pegboard Test, Minnesota Manual Dexterity Test) evaluation parameters will be applied before, immediately after and 15 minutes after each exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Female-male gender
* Not exercising regularly for the last 6 months
* Participated in the study voluntarily
* Individuals without glasses or contact lenses

Exclusion Criteria:

* BMI>30
* Individuals with a self-reported history of psychiatric, neurological, cardiovascular or pulmonary disease
* Individuals with orthopedic pathology
* Individuals with musculoskeletal dysfunction

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-12-25 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
ROM Measurement | 10 minutes
  ROM measurement will be applied by including both extremities of the participants Shoulder flexion and abduction, elbow flexion and extension while the subjects were in the supine position; While in the sitting position, forearm supination and pronation, wrist flexion and extension were evaluated respectively. Measurements were made with a universal goniometer; It was repeated three times and average values were taken as basis. The results were evaluated in degrees.
Muscle Strength Measurements | 15 minutes
  Measurements will be made with participants in a sitting position. The strength of the shoulder flexor, shoulder abductor, elbow extensor, elbow flexor muscles, forearm supination, pronation muscles, wrist extensor, and wrist flexor muscles will be checked. 'LaFayette' brand digital hand dynamometer was used to evaluate muscle strength. Muscle testing in each region was repeated three times for the right and left extremities. The best values of the right and left sides were noted. Results were evaluated in lbs.
Grip Force Measurement (Pinchmeter, Jamar hand dynamometer) | 5 minutes
  The measurement will be taken in a sitting position, with the shoulder in adduction and neutral rotation, the elbow in 90 degrees flexion, the forearm in mid-rotation and support, and the wrist in neutral. According to the test procedure, 3 measurements will be made with one-minute intervals between each measurement for hand grip strength and the averages will be recorded.The results were evaluated in kg.
Nelson Hand Reaction Test (Ruler Drop Test) | 5 minutes
  For the test, the person's dominant hand will be evaluated. The person will be asked to sit with the elbow flexed at 90 degrees and the dominant hand in a neutral position, with the forearm supported on the table. The practitioner will hold the ruler between the subject's thumb and index finger and the tips of the thumb and forefinger should be 8-10 cm ahead of the table edge and the upper parts of the thumb and forefinger should be parallel to each other. During the test, the person will be asked to look at the middle point of the ruler when the ruler is released and to catch the ruler between the thumb and index fingers. The score will be recorded by reading the line at the top of the thumb as soon as the person holds the ruler. Measurements will be repeated three times and averaged for data analysis.
Purdue Pegboard Test | 5 minutes
  The test includes a test board with 2 parallel columns and a total of 50 holes, and a platform with 4 compartments where nails, washers, and nuts are located. During the start of the test, participants will be asked to start via a verbal command while timing is kept on the stopwatch. The test consists of four subsets. Subjects will be asked to put the pegs into the holes within 30 seconds, first with the dominant hand, then with the non-dominant hand, then with both hands. In the final set, subjects will be given 1 minute to assemble a nail, a washer, a nut, and finally another washer with alternating hands, starting with the dominant hand. Each set will be repeated three times to obtain an average. Test scores will be calculated based on the number of holes filled or parts joined based on the test subset.
Minnesota Manual Dexterity Test | 5 minutes
  Participants will be asked to place 60 round cylindrical boxes in the Minnesota dexterity test protocol from right to left and from left to right against time. All participants will be asked to complete the test with the right and then the left hand, and their times will be recorded by keeping a stopwatch.

SECONDARY OUTCOMES:
Arm Ergometer | 25 minutes
  Exercise intensity will determined by the target heart rate method. Exercise intensity will be apply at 60%, 70%, 80% of the maximum heart rate at least 24 hours apart. The maximum heart rate will be determined by the 200-age formula. Exercises will be performed with an arm ergometer. Participants will asked not to do intense exercise within 12 hours before each test, stop consuming alcohol and caffeine, and to be hungry for 3 hours. The tests will repeat at the same time with a maximum deviation of 1 hour on 3 different days. Participants in the study will warm up for 5 minutes. After the warm-up, the load will be increased and the 20-minute training protocol will start. When the participants reach the desired heart rate range, 20 minutes will be completed. In total, participants will be warmed up for 5 minutes and exercised for 20 minutes. The participants will be taken directly to the tests without cooling down.

CONTACTS AND LOCATIONS:
Overall Officials: Esra PEHLİVAN, Assoc.Prof, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Saglik Bilimleri Universitesi, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No